CLINICAL TRIAL: NCT02542124
Title: A Single Arm, Open-Label Study To Evaluate The Safety, Tolerability And Preliminary Efficacy Of NM-IL-12 (rHuIL-12) In Patients With Cutaneous T Cell Lymphoma (CTCL) Undergoing Low Dose Total Skin Electron Beam Therapy (TSEBT)
Brief Title: NM-IL-12 in Cutaneous T-Cell Lymphoma (CTCL) Undergoing Total Skin Electron Beam Therapy (TSEBT)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neumedicines Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM-ONC-001; 1R44CA192576-01 (NIH)
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Cutaneous T Cell Lymphoma (CTCL); Mycosis Fungoides; Sézary Syndrome
Keywords: CTCL; Total Skin Electron Beam Therapy (TSEBT); Mycosis fungoides; Sézary syndrome; recombinant human Interleukin-12 (rHuIL-12); T Cell
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NM-IL-12 and TSEBT (Experimental): TSEBT and subcutaneous doses of NM-IL-12
  Interventions: Biological: NM-IL-12 and TSEBT

INTERVENTIONS:
Biological: NM-IL-12 and TSEBT — The LD-TSEBT treatment will start on Day 1 of the study. NM-IL-12 will be administered subcutaneously.
  Other Names: HemaMax, rHu-IL12, LD-TSEBT

SUMMARY:
In the proposed study, NM-IL-12 will be evaluated as immunotherapy to increase antitumor efficacy against CTCL, while reducing skin-related toxicity, when combined with low-dose TSEBT therapy. Determination of the maximum tolerated dose (MTD) for NM-IL-12 is not planned in this study, rather, a pre-defined starting dose will be explored; this dose is based on two safety and tolerability studies of NM-IL-12 in healthy volunteers.

DETAILED DESCRIPTION:
This is a single arm, open-label, non-randomized study with NM-IL-12 dosed in combination with low dose TSEBT in CTCL patients. This study is planned to be conducted in 10 patients, 18 years or older in age, undergoing low dose TSEBT of 12 Gy over a 3-week period.

The study will initially enroll 4 patients and then will be expanded to enroll 6 additional patients (total 10 patients) depending on the presence or absence of Dose Modifying Criteria (DMC). Decision whether to de-escalate will be made after first 4 patients are followed up for 28 days from the first dose of NM-IL-12.

Safety monitoring will continue throughout the whole period of drug administration and the treatment will be discontinued if intolerable toxicity or disease progression occurs during this period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Biopsy-confirmed CD4+ mycosis fungoides or Sézary syndrome, stage IB to IIIB
3. The patient is eligible for TSEBT
4. Eastern Cooperative Oncology Group (ECOG) of ≤ 2.
5. Adequate bone marrow function: WBC > 2000/μL; platelet count > 75,000/μL; Neutrophil count > 1000/μL, without use of colony stimulating factors (CSF).
6. Required washout period for prior therapies Topical therapy: 2 weeks

   * Phototherapy (PUVA): 4 weeks
   * Local Skin Radiation Therapy (< 10% skin surface): 4 weeks
   * Retinoids: 4 weeks
   * Interferons: 4 weeks
   * Low dose methotrexate: 4 weeks
   * HDAC inhibitors: 8 weeks
7. Women of child-bearing potential must have negative serum pregnancy test and use accepted highly effective methods of birth control throughout the study and for 90 days after dosing and must agree to use effective contraception.
8. Male patients must be willing to use an appropriate method of contraception (e.g., condoms) or abstain from sexual intercourse and inform any sexual partners that they must also use a reliable method of contraception during the study and for 90 days after dosing.
9. Adequate hepatic function: bilirubin ≤1.5 x upper limit of normal (ULN), AST ≤2.5 x ULN, ALT ≤2.5 x ULN, alkaline phosphatase (liver fraction) ≤2.5 x ULN
10. Adequate renal function: creatinine ≤1.5 x ULN
11. Ability to comply with the treatment schedule

Exclusion Criteria:

1. Biopsy confirmed CD8+ CTCL histology
2. Large cell transformation
3. Prior systemic use of any immunosuppressive chemotherapy (except low dose methotrexate) and/or monoclonal antibody treatment for CTCL
4. Prior courses of TSEBT (Note: localized skin-directed radiotherapy is allowed if administered at least 4 weeks prior to initiation on study).
5. Concomitant use of any anti-cancer therapy or immune modifier.
6. Prior allogeneic hematopoietic cell transplant.
7. Any ongoing infection whether receiving or not receiving antibiotics or have received intravenous antibiotics, antiviral, or antifungal agents within 2 weeks prior to the start of the study drug.
8. Known history of human immunodeficiency virus (HIV), hepatitis B or C
9. For women on estrogen based contraceptives, family history of venous thromboembolism (VTE) and/or risk factors predisposing for VTE and other medical conditions known to be associated with VTE.
10. History of prior malignancy with the exception of cervical intraepithelial neoplasia, non-melanoma skin cancer, and adequately treated localized prostate carcinoma (PSA <1.0). Patients with a history of other malignancies must have undergone potentially curative therapy and have no evidence of that disease for five years
11. Uncontrolled intercurrent illness, condition, or circumstances that could limit compliance with the study, including, but not limited to the following: acute or chronic graft versus host disease, uncontrolled diabetes mellitus or hypertension, or psychiatric conditions
12. Any other medical issue, including laboratory abnormalities, deemed by the Investigator to be likely to interfere with patient participation
13. Unresolved toxicity from previous anticancer therapy or incomplete recovery from surgery
14. Major surgery within 12 weeks of enrolment
15. Medically significant cardiac event or unstable cardiovascular function defined as:

    * Symptomatic ischemia, unstable angina pectoris
    * Uncontrolled clinically significant cardiac arrhythmia
    * Symptomatic heart failure NYHA Class ≥ 3
    * Myocardial infarction or cardiac surgery within 6 months prior to enrollment
16. Cerebrovascular event (transient ischemic attack, stroke or CNS bleeding) within the last 12 months.
17. Major bleeding within the last 6 months.
18. Use of any investigational agents within 30 days prior to enrollment and for the duration of the study
19. Pregnant or lactating
20. Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated on the basis of the following parameters (Vital signs, physical examination,Toxicity according to the NCI CTCAE, Immunogenicity evaluated by the presence of anti-drug antibody) : | 107 weeks
  General safety: Vital signs (temperature, blood pressure, pulse rate, respiratory rate) and physical examination.
  Toxicity according to the NCI CTCAE (v4.03) for AEs and clinical laboratory profile; AEs will be collected in all patients who received at least one dose of NM-IL-12 and up to four weeks post last NM-IL-12 dose.
  Immunogenicity of NM-IL-12 will be evaluated by the presence of anti-drug antibody (ADA)

SECONDARY OUTCOMES:
Clinical Response measured by a modified severity-weighted assessment tool (mSWAT) | 107 weeks
  Exploratory skin clinical responses measured by a modified severity-weighted assessment tool (mSWAT)
Progression free survival | 107 weeks
  Progression free survival based on every 4 week follow up after the monthly dose until one of the events below occurs first:
  * Progressive disease is documented
  * Another treatment for CTCL is administered (topical or systemic)
  * 107 weeks are completed after the patient's first dose of NM-IL-12

CONTACTS AND LOCATIONS:
Overall Officials: Youn H Kim, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford Cancer Center, Stanford, California
  - Columbia University Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gokhale MS, Vainstein V, Tom J, Thomas S, Lawrence CE, Gluzman-Poltorak Z, Siebers N, Basile LA. Single low-dose rHuIL-12 safely triggers multilineage hematopoietic and immune-mediated effects. Exp Hematol Oncol. 2014 Apr 11;3(1):11. doi: 10.1186/2162-3619-3-11. PMID 24725395
- [Background] Gluzman-Poltorak Z, Vainstein V, Basile LA. Recombinant interleukin-12, but not granulocyte-colony stimulating factor, improves survival in lethally irradiated nonhuman primates in the absence of supportive care: evidence for the development of a frontline radiation medical countermeasure. Am J Hematol. 2014 Sep;89(9):868-73. doi: 10.1002/ajh.23770. Epub 2014 Jun 19. PMID 24852354
- [Background] Gluzman-Poltorak Z, Mendonca SR, Vainstein V, Kha H, Basile LA. Randomized comparison of single dose of recombinant human IL-12 versus placebo for restoration of hematopoiesis and improved survival in rhesus monkeys exposed to lethal radiation. J Hematol Oncol. 2014 Apr 6;7:31. doi: 10.1186/1756-8722-7-31. PMID 24708888
- [Background] Basile LA, Ellefson D, Gluzman-Poltorak Z, Junes-Gill K, Mar V, Mendonca S, Miller JD, Tom J, Trinh A, Gallaher TK. HemaMax, a recombinant human interleukin-12, is a potent mitigator of acute radiation injury in mice and non-human primates. PLoS One. 2012;7(2):e30434. doi: 10.1371/journal.pone.0030434. Epub 2012 Feb 24. PMID 22383962
- [Background] Rook AH, Wood GS, Yoo EK, Elenitsas R, Kao DM, Sherman ML, Witmer WK, Rockwell KA, Shane RB, Lessin SR, Vonderheid EC. Interleukin-12 therapy of cutaneous T-cell lymphoma induces lesion regression and cytotoxic T-cell responses. Blood. 1999 Aug 1;94(3):902-8. PMID 10419880
- See also: Single Low-dose rHuIL-12 Safely Triggers Multilineage Hematopoietic and Immune-mediated Effects. — http://www.ehoonline.org/content/3/1/11